CLINICAL TRIAL: NCT06521164
Title: Usability of Pericardial Flushing with the Haermonics Pure System After Cardiac Surgery
Acronym: USEPURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haermonics BV (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-2024-0047
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Surgical Blood Loss; Surgical Complication
Keywords: cardiac surgery; therapeutic irrigation; postoperative bleeding; chest tubes; Haermonics Pure System
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study subjects (Other): 1-arm study
  Interventions: Device: Haermonics Pure system

INTERVENTIONS:
Device: Haermonics Pure system — pericardial flushing with Haermonics Pure system

SUMMARY:
The goal of this clinical trial is to evaluate the usability of the Haermonics Pure system in patients undergoing a cardiac surgery procedure with the use of cardiopulmonary bypass.

All measurements and interventions are standard of care, except pericardial flushing with the Haermonics Pure system.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center clinical investigation of adult patients undergoing cardiac surgery. Safety and efficacy of CPPF, with and without the device, has been established in comparison with standard drainage. Therefore, this study is designed primarily to establish the usability of the device and its accessories, not requiring randomization against a control group.

Because the Haermonics Pure system and its accessories are used directly after surgery for several hours up to several days until drain removal before being discharged from the hospital, it is sufficient to follow patients until discharge from the cardiac surgery department. For patients with a prolonged hospitalization because of postoperative complications, it is considered sufficient to follow patients for 2 weeks after surgery because the impact of a pericardial flushing and postoperative drainage on outcomes is critical within the immediate postoperative period but limited beyond the time that the drains are removed. For device-related adverse events, follow-up will continue until the event is considered resolved or the patient is discharged.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18yrs and weight ≥40kg) undergoing cardiothoracic surgery (CABG and/or valve surgery, elective aortic surgery, Bentall procedure, ascending aorto/aortic arch replacement) with the use of cardiopulmonary bypass
2. Patient has been informed of the nature of the clinical investigation and is willing and able to give written informed consent for investigation participation

Exclusion Criteria:

1. Euroscore II > 20%
2. Emergent procedures
3. Complication during surgery which is life threatening and/or requires another surgical intervention
4. Minimal invasive cardiac surgery procedures (e.g. minithoracotomy and hemisternotomy)
5. Thoraco-abdominal surgery, or intraoperative injury to the diaphragm leading to an open connection between the thoracic and abdominal cavity
6. Participation in any study involving an investigational drug or device
7. Patient is pregnant or nursing
8. Inability to understand study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Usability to evaluate user satisfaction and functionality of all use aspects of the Haermonics Pure system within 65 patients by using a user questionnaire. | for all users at the end of the study, after enrollment of 65 patients, after approximately 5 months after the start of the study.
  For each user, questions will be asked about the common use of the Hearmonics Pure system using a 0-10 Numeric Rating Scale.
Usability to evaluate user satisfaction and functionality of all use aspects of the Haermonics Pure system within 65 patients by using a user questionnaire. | for all users at the end of the study, after enrollment of 65 patients, after approximately 5 months after the start of the study.
  For each user, questions will be asked about the use of the Hearmonics Pure system in comparison with standard practice, with option 1 Hearmonics Pure system being better, with option 2 no difference, with option 3 standard of care being better.
Usability to evaluate user satisfaction and functionality of all use aspects of the Haermonics Pure system within 65 patients by using a user questionnaire. | for all users at the end of the study, after enrollment of 65 patients, after approximately 5 months after the start of the study.
  For each user, questions will be asked about the common use of the Hearmonics Pure system using the System Usability Scale (SUS). It is comprised of 10 questions that should be answered on a 5-point Likert scale.

SECONDARY OUTCOMES:
Safety: Rate of device-related events up to discharge | From enrollment up to discharge or up to 2 weeks after surgery, whichever came first
  Descriptive statistics
Usability to evaluate user satisfaction and functionality of all use aspects of the Haermonics Pure system within 65 patients by using a user questionnaire. | For each user at each step for each patient trough study completion, which is expected to be around 3 times a week during approximately 5 months.
  Used by different user groups in different hospital settings when using the different components of the Haermonics Pure system for the different functionalities. User satisfaction is measured with a user questionaire, containing questions with a scale from 1-4, with 1: very unsatisfied, 2: unsatified; 3 satisfied; 4 very satisfied.
Safety: Rate of SAEs up to discharge | From enrollment up to discharge or up to 2 weeks after surgery, whichever came first
  Relationship with the device will be determined for all SAEs. All events of reoperations, pericardiocetesis and pleurcentesis are considered to be SAEs.
Efficacy: Drain fluid output 8 hours after start treatment (with sternum closed). | start treatment (flushing) up to 8 hours after start treatment (flushing).
  Total amount of fluid output, comparing this with the historical control established in the previous FLUID trial.
Technical Efficacy: Number of device deficiencies leading to permanently stopping the treatment for each patient, 65 patients in total | start treatment (flushing) up to removal of drains, which is typically 12-24 hours after surgery
  Device deficiencies will be recorded, including the description of the technical issue.
Efficacy: Occurance of drain occlusion | start treatment (flushing) up to removal of drains, which is typically 12-24 hours after surgery
  Having to permanently stop flushing as a result of retained fluid and no chest tube output. Patients with chest tube output until flushing is terminated and without retention that is not produced after flushing is terminated will by default not have occluded drains. It will be collected how many times the infusion was paused and/ or stopped due to fluid retention for each patient.

IPD SHARING:
Plan to Share IPD: No